CLINICAL TRIAL: NCT02320630
Title: The Efficacy, Safety and Cost-effectiveness of Hydroxychloroquine, Sulfasalazine, Methotrexate Triple Therapy in Preventing Relapse Among Patients With Rheumatoid Arthritis Achieving Clinical Remission or Low Disease Activity
Brief Title: Combination Therapy Prevents the Relapse of RA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Peking University Third Hospital (Other); Beijing Hospital (Other Government); Beijing Jishuitan Hospital (Other); Peking University Shougang Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Zhuoli Zhang, Rheumatology and Immunology Department, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCRP201305
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Recurrence (Disease Attribute)
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Maintenance treatment group
  Interventions: Drug: Entanercept; Drug: MTX
- B (Experimental): Combination treatment group
  Interventions: Drug: Entanercept; Drug: HCQ; Drug: MTX
- C (Experimental): Single drug group
  Interventions: Drug: Entanercept; Drug: MTX

INTERVENTIONS:
Drug: Entanercept — Both Entanercept and MTX were given to patients for 60weeks (Week0-Week60).
  Other Names: MTX
Drug: HCQ — Combination of HCQ+SSZ+MTX were given to patients for 60weeks (Week0-Week60).Entanercept was given to patients for 12 weeks (Week0-Week12).
  Other Names: SSZ; MTX; TFP
  Arms: B
Drug: MTX — MTX was given to patients for 60weeks (Week0-Week60). Entanercept was given to patients for 12 weeks (Week0-Week12).
  Other Names: Entanercept

SUMMARY:
This trial aims to compare the cost effective and effect of preventing recurrence by different treatment of TFP and HCQ combined SSZ for remittent RA.

DETAILED DESCRIPTION:
patients were divided into 3groups: Group A:TFP+MTX (week0-week60) Group B:TFP+MTX+HCQ+SSZ(week0-week12) and then MTX+HCQ+SSZ(week13-week60) Group C:TFP+MTX (week0-week12) and then MTX (week13-week60)

ELIGIBILITY:
Inclusion Criteria:

* Fulfill 2010 EULAR/ACR RA dignose criteria
* Age18-70 years old
* Have been teated regularly for 3 months
* Disease duration > 6months
* DAS28>3.2

Exclusion Criteria:

* Received surgical operation in 8 weeks
* Received other biological agent (eg. rituximab, anti-TNF agents, anti-IL6 agents)in 6 months;
* Injection of steroid in 4 weeks
* Coexisting with other CTD except for SS
* With severe and not controled cardiac vescular disease, neurological disease, pulmonary disease (including COPD and ILD), renal disease, liver disease, endocrine disease and Gastric Intestinal Disease
* With not controled diseases including asthma, IBD and psoriasis needing oral or injection of steroid
* Active infection with T>38℃. Patients need admitted into hospital or biotics injection in 4 weeks or need oral biotics in 2 weeks
* Malignant history.
* Serum creatinine >130 µmol/L
* AST/ALT higher than 2 times upper level
* platelet count<100 x 109/L，or white blood count<3 x 109/L
* Interstitail lung disease: Chest X Ray
* Hands X Ray ACR radiology staging shows IV stage RA
* Pregnancy or planing to pregnant in 2 years or suckling period women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the rate of recurrence | 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology and Immunology Department,Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao J, Zhou W, Wu Y, Yan X, Yang L, Zhang Z. Efficacy, safety, and cost-effectiveness of triple therapy in preventing relapse in rheumatoid arthritis: A randomized controlled trial (ESCoRT study). Chin Med J (Engl). 2022 Sep 20;135(18):2200-2209. doi: 10.1097/CM9.0000000000002336. PMID 36525606
- [Derived] Zhao J, Zhou W, Wu Y, Ji P, Yang L, Yan X, Zhang Z. The efficacy, safety and cost-effectiveness of hydroxychloroquine, sulfasalazine, methotrexate triple therapy in preventing relapse among patients with rheumatoid arthritis achieving clinical remission or low disease activity: the study protocol of a randomized controlled clinical Trial (ESCoRT study). BMC Med Inform Decis Mak. 2021 Mar 4;21(1):83. doi: 10.1186/s12911-021-01449-2. PMID 33663487
- [Derived] Fan Y, Yang X, Zhao J, Sun X, Xie W, Huang Y, Li G, Hao Y, Zhang Z. Cysteine-rich 61 (Cyr61): a biomarker reflecting disease activity in rheumatoid arthritis. Arthritis Res Ther. 2019 May 21;21(1):123. doi: 10.1186/s13075-019-1906-y. PMID 31113467